CLINICAL TRIAL: NCT01187732
Title: WASHING WITHOUT WATER Cost-effectiveness of a Rapidly Spreading Nursing Intervention om Bedridden Patients'
Brief Title: Washing Without Water: Cost-effectiveness of a Rapidly Spreading Nursing Intervention in Bedridden Patients'
Acronym: WWW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Betsie van Gaal (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor-Investigator, Betsie van Gaal, PhD, Radboud University Medical Center
Organization: Radboud University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 80-82310-97-1074
Record Dates: First submitted 2010-08-23; First posted 2010-08-24 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Skin Disease
Keywords: skin damage; intertrigo; dermatitis; erythema; aggression; body Wipes; soaps; no rinse; cost effectiveness; nursing home residents; nurse
MeSH Terms: conditions — Skin Diseases; Intertrigo; Dermatitis; Erythema; Aggression | interventions — Therapeutic Irrigation; Hydrotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Washing without water (Experimental): The experimental intervention is 'washing without water' and consists of disposable washing cloths made of a mix of soft synthetic fibers, saturated with a no rinse, quickly vaporizing skin cleaning and caring lotion.
  Interventions: Device: Washing without water
- Traditional soap and water bath (Active Comparator): The control intervention is the traditional bathing assistance as performed in care dependent patients by using tap water, a bowl, towels, washcloths and soap.
  Interventions: Device: Washing without water

INTERVENTIONS:
Device: Washing without water — The experimental intervention is 'washing without water' and consists of disposable washing cloths made of a mix of soft synthetic fibers, saturated with a no rinse, quickly vaporizing skin cleaning and caring lotion.
  Other Names: bag baths; disposable washing cloths

SUMMARY:
The purpose of this study is to compare the traditional bed bath with 'washing without water' on

* 1) effects on skin integrity
* 2) patient and nurse satisfaction and 3) costs. In a cluster randomized trial we will randomize 50 nursing home wards (576 patients) to 'washing without water' or traditional bed baths. Bathing regimens are continued for six weeks.

Whereas effects on skin damage are not likely to be specific for setting, these results can be generalized to other patient groups.

DETAILED DESCRIPTION:
RAPID IMPLEMENTATION of new interventions while cost-effectiveness and acceptability for patients and care providers are unclear, is never desirable. 'Washing without water' is such an intervention.

The traditional bed bath is executed by using tap water, towels, washcloths and soap. As an alternative, 'WASHING WITHOUT WATER' was recently introduced in the Netherlands. This concept consists of disposable washcloths made of a mix of soft synthetic fibers, saturated with a no rinse, quickly vaporizing skin cleaning and caring lotion. 'WASHING WITHOUT WATER' can be used with all patients who need bathing assistance, especially when taking a shower or sitting in a hot tub is not possible.

However, while several claims are made about the positive effects of 'washing without water' as compared to traditional bathing, EVIDENCE IS LACKING. Also, 'washing without water' is CONTROVERSIAL. While some are eager to adopt the new concept, others see it as 'efficiency gone loose' and denying patients one of the most basic elements of care: a proper bath. This study therefore addresses the cost effectiveness of 'washing without water' in bedridden patients.

ELIGIBILITY:
Inclusion Criteria:

* long stay psychogeriatric nursing home residents
* long stay somatic nursing home residents
* 100 randomly selected nurses from the participating nursing home wards

Exclusion Criteria:

-

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2011-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
the primary outcome is prevalence of care associated skin damage | 6 weeks
  Skin damage is defined as intertrigo, dermatitis and/or other erythema on skin areas which were not exposed to pressure directly before observation.

SECONDARY OUTCOMES:
Patient and nurse satisfaction with bathing technique | 6 weeks
  * patient perceived discomfort during bathing
  * nurse perceived work load
  * observed bathing quality
Cost bathing | 6 weeks
  Bathing and skin damage associated costs will be calculated from the costs of bathing and skin care associated staff time and the materials used.

CONTACTS AND LOCATIONS:
Overall Officials: Theo van Achterberg, PhD, Study Chair — Radboud university medical center; IQ healthcare
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schoonhoven L, van Gaal BG, Teerenstra S, Adang E, van der Vleuten C, van Achterberg T. Cost-consequence analysis of "washing without water" for nursing home residents: a cluster randomized trial. Int J Nurs Stud. 2015 Jan;52(1):112-20. doi: 10.1016/j.ijnurstu.2014.08.001. Epub 2014 Aug 10. PMID 25173772